CLINICAL TRIAL: NCT01613716
Title: Ozurdex for Diabetic Macular Edema Treated With Pars Plana vitrEctomy and Membrane RemovAl (OPERA Study)
Acronym: OPERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Sunil Srivastava, PI, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115200
Record Dates: First submitted 2012-06-05; First posted 2012-06-07 (Estimated); Results first posted 2018-05-16 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-04

CONDITIONS: Diabetic Macular Edema; Epiretinal Membrane
Keywords: Diabetes; Macular Edema; Epiretinal Membrane; Vitrectomy
MeSH Terms: conditions — Epiretinal Membrane; Diabetes Mellitus; Macular Edema | interventions — Calcium Dobesilate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ozurdex (Experimental): Subjects will receive Ozurdex injections and will be monitored for macular edema.
  Interventions: Drug: Ozurdex

INTERVENTIONS:
Drug: Ozurdex — Ozurdex .7 mg injected into the treated eye
  Other Names: Dexamethasone

SUMMARY:
This study will examine the use of the dexamethasone implant (Ozurdex) in patients with macular edema associated with an epiretinal or preretinal membrane requiring surgical intervention. After the surgery is performed (pars plana vitrectomy), an Ozurdex implant will be placed in the eye. Patients will be followed for 1 year.

DETAILED DESCRIPTION:
The purpose of this study to examine the use of Ozurdex in patients who are undergoing pars plana vitrectomy for macular edema due to preretinal membranes. Specifically, we will examine its effect on macular edema (measured by OCT), and visual recovery (measured by visual acuity). We will examine its use in patients who underwent pars plana vitrectomy for macular edema with associated taut membrane. This will be a prospective pilot study with patients to receive an Ozurdex implant at the time of vitrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are undergoing pars plana vitrectomy for:

   * Epiretinal membrane/vitreomacular traction or
   * Diabetic macular edema
2. Patients with macular edema as measured by OCT (at least 250 um central subfoveal thickness)
3. Informed consent requirements: All study subjects must agree to participate in the study and provide written informed consent, which will be written in English.
4. Age between 18-85 years old

Exclusion Criteria:

1. Age < 18 years or > 85 years
2. History of macular edema due to diseases other than those in the inclusion criteria in the study eye

   * History of active inflammatory eye disease (uveitis) (within 3 months)
   * History of ocular malignancy and/or ocular/orbital irradiation
   * History of recent retinal vein occlusion (within 6 months)
   * History of neovascular age-related macular degeneration or choroidal neovascular membrane [
   * History of juxtafoveal telangiectasia
   * History of Coat's disease
   * History central serous choroidoretinopathy
   * History of previous infectious retinitis (toxoplasmosis, acute retinal necrosis, tuberculosis, etc)
3. Patients with a history of intraocular infection in the study eye (i.e. viral retinitis, endophthalmitis)
4. Patients who are cognitively impaired or those who are unable to provide informed written consent
5. Patients with a history of glaucoma in the study eye (defined as increased cup to disc ratio with associated nerve damage. Patients with ocular hypertension controlled by topical glaucoma drops (maximum 3) will not be excluded).
6. Patient with recent intravitreal injections of steroids or anti-VEGF medications in the study eye (within past 4 weeks).
7. Patients with recent periocular steroid injection (within past 4 weeks) in the study eye
8. Patients on topical NSAIDS drops (patient will be eligible if they discontinue use of topical NSAIDs at time of study enrollment) in the study eye

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Srivastava, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cole Eye Institute, Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ozurdex
Started | 30
Completed | 23
Not Completed | 7
Not completed — screen failures | 3
Not completed — Lost to Follow-up | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ozurdex
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 61.63 [37 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Central Retinal Thickness
Description: At 3 months, central retinal thickness as measured by optical coherence tomography will be measured
Time Frame: 3 months
Population: Optical Coherence Tomography was collected at 3 months. 22 of the patients were seen at month 3.
Measure: Median (Full Range); unit: micrometers
Arm/Group | Ozurdex
Number analyzed (Participants) | 22
micrometers | 350 [208 to 483]

2. Primary Outcome: Visual Acuity
Description: ETDRS visual acuity will be measured at 3 months. Visual function of the study eye was assessed using the ETDRS protocol, which is a widely accepted international standard. A higher letter score represents better functioning.
Time Frame: 3 months
Population: 23 of the participants were able to come in for their 3 month appointment per protocol
Measure: Median (Full Range); unit: ETDRS
Arm/Group | Ozurdex
Number analyzed (Participants) | 23
ETDRS | 56 [0 to 85]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from point of screening until their last visit at 12 months.
Arm/Group | Ozurdex
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 7/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex (N=30)
Persistent Corneal Epithelial Defect (Eye disorders) | 1 (1) — Patient had a persistent corneal defect after vitrectomy surgery and implantation of Ozurdex. Subsequently healed.
Area of tractional retinal detachment versus retinoschisis surgery eye (Eye disorders) | 1 (1) — Patient had an are of possible tractional retinal detachment versus retinoschisis noted throughout the surgery after vitrectomy surgery.
Peptic ulcers-hospitalized for stomach pain (Gastrointestinal disorders) | 1 (1) — Patient had a bout of stomach and was hospitalized and diagnosed with peptic ulcers.
Root canal infection (Infections and infestations) | 1 (1) — Patient had a root canal and developed an infection afterwards
Removal of basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Patient had a biopsy of the nose that was subsequently diagnosed as a basal cell carcinoma
Ozurdex placment on fovea (Eye disorders) | 1 (1) — After placement of Ozurdex it adhered to the fovea, requiring a second surgery where it went back into the normal position.
Myocardial infarction (Cardiac disorders) | 1 (1) — Patient subsequently underwent a CABG procedure, had a previous history of cardiac issues.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ozurdex (N=30)
Increase in cataract surgical eye (Eye disorders) | 2 (2) — Increase in cataract in the surgical eye
Increase in cataract fellow eye (Eye disorders) | 6 (6) — Increase in cataract surgery fellow eye
Increase in intraocular pressure (Eye disorders) | 7 (7) — Increase in intraocular pressure
Worsening of diabetic disease fellow eye (Eye disorders) | 8 (19) — Worsening of diabetic eye disease or cystoid macular edema
Motor vehicle accident (Injury, poisoning and procedural complications) | 2 (2) — Patient was involved motor vehicle collusion no hospitalizations
worsening of posterior capsular opacity (Eye disorders) | 3 (3) — Worsening of posterior capsular opacity study eye
worsening of posterior capsular opacity fellow eye (Eye disorders) | 1 (1) — As described above
respiratory flu (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory flu
Dental infection (Infections and infestations) | 1 (1) — Infection after dental procedure
Poison Ivy rash (Skin and subcutaneous tissue disorders) | 1 (1) — Was treated in the emergency room for poison ivy.
Tachycardia (Cardiac disorders) | 1 (1) — found during a sleep study during a cardiology visit.
broken patella (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchitis (Reproductive system and breast disorders) | 1 (1)
increased cystoid macular edema study eye (Eye disorders) | 5 (7)
Transient Ischemic Avent (Nervous system disorders) | 1 (1) — Patient had history of previous TIAs
Epithelial defect study eye (Eye disorders) | 4 (4) — Patient had reported epithelial defect after vitrectomy surgery.
Increased itching both eyes (Eye disorders) | 4 (4)
Increase in pain study eye (Eye disorders) | 2 (2) — Patient noted increased pain in surgical eye
Increased diabetic retinopathy study eye (Eye disorders) | 1 (1)
Increase of dryness of the eyes (Eye disorders) | 2 (2)
Trouble breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — patient was diagnosed with pneumonia
Cartoid blockage (Cardiac disorders) | 1 (1) — Patient had previous history of blockage was scheduled for outpatient stent
loss of vision fellow eye (Eye disorders) | 1 (1) — Patient reported decrease vision fellow eye
small choroidal study eye (Eye disorders) | 1 (1) — Choroidal was found postoperatively from vitrectomy surgery.
Vitreous hemorrhage study eye (Eye disorders) | 2 (2) — Patient had a vitreous hemorrhage of study eye
Syncope after injection (General disorders) | 1 (1) — patient had syncope episode after protocol injection of ozurdex
Trouble reading (Eye disorders) | 1 (1) — Patient reported difficulty with reading both eyes
Nausea, vomiting diarrhea,dehydration (Injury, poisoning and procedural complications) | 1 (1) — Went to the emergency room the night of surgery with complications of anesthesia from vitrectomy surgery- was not admitted
Worsening of Parkinson's tremors (Nervous system disorders) | 1 (1) — Patient had past medical history of Parkinson's
Sarcoidosis Flare (Immune system disorders) | 1 (2) — Patient had a flare of previously diagnosed sarcoidosis
Foreign body sensation of eyes (Eye disorders) | 1 (1) — Patient reported feeling like something was in their eyes and irritating it- nothing was found in their eyes.
Injury to hip an back (Injury, poisoning and procedural complications) | 1 (1) — Patient had a work related injury requiring physical therapy
Diarrhea (Gastrointestinal disorders) | 1 (1) — Patient reported diarrhea, did not seek medical attention
Subconjunctival hemorrhage fellow eye (Eye disorders) | 1 (1)
Digestion issues (Gastrointestinal disorders) | 1 (2) — Patient had reported digestion issue later diagnosed with GERD
Sinus infection (Infections and infestations) | 2 (2) — Reported sinus infections
Increased floaters fellow eye (Eye disorders) | 2 (2)
Decreased television vision fellow eye (Eye disorders) | 1 (1)
Glare with vision at night (Eye disorders) | 1 (1)
Tearing in both eyes (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No